CLINICAL TRIAL: NCT05601206
Title: Collaborative Care Intervention for Cancer Patients and Their Family Caregivers -LITE
Acronym: CARES-Lite
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Care coordinators graduated
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jennifer Steel, Director and Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY22050018
Record Dates: First submitted 2022-08-29; First posted 2022-11-01 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Depression; Fatigue; Pain; Sleep
Keywords: Cancer Depression Fatigue Pain
MeSH Terms: conditions — Neoplasms; Depression; Fatigue; Pain | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepped collaborative care intervention (Experimental): The 'Stepped Collaborative Care Intervention' includes at least biweekly contact from a care coordinator by phone and face to face visits occurring approximately every 2 months, and 24 hour 7 day a week access to a website that was specifically designed during the pilot study for advanced cancer patients from socioeconomically disadvantaged backgrounds.
  Interventions: Behavioral: Stepped collaborative care intervention
- Enhanced Usual Care (Active Comparator): Patients randomized to the 'Enhanced Usual Care' arm receive their usual care from their medical team. However, if the patient scores in the clinical range on one or more of the three symptoms s/he will receive education about the symptom and be referred to the appropriate health care provider for further treatment in their community. The care coordinator will follow up with the patient after 3 weeks to assess barriers to treatment and assist further with accessing treatment if needed.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Stepped collaborative care intervention — Using website that was specifically designed for advanced cancer patient, collaborative with treatment from health professional
  Other Names: Treatment
  Arms: Stepped collaborative care intervention
Behavioral: Enhanced Usual Care — Usual care from health providers
  Other Names: Control
  Arms: Enhanced Usual Care

SUMMARY:
To test the efficacy of a web-based stepped collaborative care intervention to reduce symptoms of depression, pain, and fatigue and improve health-related quality of life (HRQL) in advanced cancer patients and to reduce stress and depression, and fewer CVD risk factors in caregivers.

DETAILED DESCRIPTION:
The intervention is designed to maintain quality of life for those in greatest need and least access to resources. This innovative and scalable web-based collaborative care intervention is expected not only to improve patients' quality of life, at the end of life, but also reduce caregiver stress and depression, and potentially health morbidity and mortality of patients and spousal and intimate partner caregivers from socioeconomically disadvantaged backgrounds. Study findings are expected to lead to research examining the dissemination and implementation of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

Biopsy and/or radiograph proven diagnosis of hepatocellular carcinoma, cholangiocarcinoma, gallbladder carcinoma or breast, ovarian, or colorectal cancer with liver metastases with a life expectancy of at least one year; age >21 years; no evidence of thought disorder, delusions, or active suicidal ideation is observed or reported.

* Caregivers:

A spouse or cohabitating intimate partner of an advanced cancer patient being evaluated the UPMC's Liver Cancer Center and age >21 years

Exclusion Criteria:

* Patients:

Age < 21 years, Lack of fluency in English, Evidence of thought disorder, delusions, hallucinations, or suicidal ideation.

* Caregivers:

Age < 21 years, Lack of fluency in English, Evidence of thought disorder, delusions, hallucinations, or suicidal ideation.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-14 (Estimated); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality | Change from baseline at 6 months
  Pittsburgh Sleep Quality Index (PSQI)
Pain Level | Change from baseline at 6 months
  Brief Pain Inventory (BPI)
Functioning | Change from baseline at 6 months
  Functional Assessment for Cancer Therapy Hepatobiliary (FACT - Hep)
Depression | Change from baseline at 6 months
  Center for Epidemiological Studies -Depression (CESD)
Stress | Change from baseline at 6 months
  Perceived Stress Scale (PSS)
Fatigue | Change from baseline at 6 months
  Functional Assessment for Cancer Therapy Fatigue (FACT - Fatigue)
Caregiver Quality of Life | Change from baseline at 6 months
  Caregiver Quality of Life Questionnaire (CQOL)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Steel, Principal Investigator — UPMC Department of Surgery
Locations (2):
- United States (2):
  - University of Pittsburgh Medical Center Montefiore Liver Cancer Center, Pittsburgh, Pennsylvania
  - University of Pittsburgh's Medical Center Montefiore Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-Identified Data may be shared with investigators who request data from the Primary Investigator
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available at the end of the study for up to one year.
Access Criteria: Appropriate investigator credentials (MD, PhD) and request, and for up to one year after study completion